CLINICAL TRIAL: NCT05775770
Title: Survey of Practices on the Management of Glycemia in Patients Hospitalized in Intensive Care Units
Brief Title: Blood Glucose Management in Intensive Care Units
Acronym: GINGER
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: French Society for Intensive Care (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-A01304-39
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Insulin Hypoglycemia; Glucose Test Site Bleeding; Hyperglycemia
Keywords: glucose control; insulin
MeSH Terms: conditions — Hyperglycemia; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Insulin — insulin therapy

SUMMARY:
The investigators propose to conduct a study of practices to describe the methods of managing glycemic control in hospitalized patients in critical care. This is a prospective multicenter observational study conducted in Intensive Medicine and Resuscitation departments in France and Belgium. The aim of this study is to carry out an inventory of the current practices of glycemia management as well as their modalities. Being one of the key points of the management, this work will have for main objective to raise the importance of the glycemic variabilities according to the methods of insulin therapies used.

ELIGIBILITY:
Inclusion Criteria:

* Patient with hyperglycaemia requiring an insulin prescription within 48 hours of admission
* Insulin therapy started less than 12 hours before inclusion of the patient in the study
* Expected duration of hospitalization greater than or equal to 48 hours

Exclusion Criteria:

* Moribund patients
* Patients admitted for ketoacidosis or hyperosmolar coma
* Patients admitted for symptomatic hypoglycaemia
* Patient requiring insulin for serum potassium correction
* Severe acute hepatocellular insufficiency
* Age < 18 years old
* Pregnant or breastfeeding women
* Patients under legal protection measures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to intensive care or intensive care.
Sampling Method: Probability Sample
Enrollment: 525 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-03-12 (Estimated); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
glycemic variability | 48 hours
  Study the impact of glycemic management protocols on the glycemic variability of patients hospitalized in intensive care

SECONDARY OUTCOMES:
adverse outcomes | 48 hours
  incidence of hypoglycaemia
Analysis of nursing workload | 48 hours
  nurse / patient ratio

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Papazian, Study Director — French Society for Intensive Care
Locations (1):
- CHU Caen, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided